CLINICAL TRIAL: NCT06158412
Title: A Single-center, Prospective, Single-arm Clinical Study of All-trans Retinoic Acid in Combination With a KPD Regimen for the Treatment of Refractory/Relapsed Multiple Myeloma (MM)
Brief Title: All-trans Retinoic Acid in Combination With a KPD Regimen for the Treatment of Refractory/Relapsed Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-08
Record Dates: First submitted 2023-11-22; First posted 2023-12-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATRA in Combination with a KPD Regimen (Experimental): All-trans Retinoic Acid plus the KPD Regimen
  Interventions: Drug: All-trans Retinoic Acid in combination with the KPD Regimen

INTERVENTIONS:
Drug: All-trans Retinoic Acid in combination with the KPD Regimen — Regimen: 1 course of treatment for 28 days until disease progression or intolerable toxicity occurs
  1. ATRA mg/m2/day in 2 oral doses for 3 days. The first dose of ATRA will be given in the morning, two days prior to carfilzomib administration.
     The last ATRA dose will be given in the evening on the day of carfilzomib administration.
  2. Proteasome inhibitor: Carfilzomib 27mg/m2 2 consecutive days per week x 3 weeks (20mg/m2 on day 1 and day 2 of cycle 1);
  3. Pomalidomide 4mg orally daily, d1-21;
  4. Dexamethasone given orally only on days 1, 8, 15, and 22 of each cycle; ≤75 years: 40 mg/day; >75 years: 20 mg/day.

SUMMARY:
To investigate the safety and efficacy of the ATRA combined with the KPD regimen in patients with refractory relapsed multiple myeloma.

DETAILED DESCRIPTION:
This is an open-label clinical trial study that aims to evaluate the efficacy (eg. Complete response, Overall Survival, Progression Free Survival) and adverse effects of Trans-Retinoic acid (ATRA) combined with the KPD regimen in patients with refractory relapsed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Subjects must have a diagnosis of multiple myeloma based on the following criteria: (1) Monoclonal plasma cells in the bone marrow in ≥10% of patients at some point in time when the presence of plasmacytoma is confirmed by disease history or biopsy. (2) Measurable disease is defined as follows: Serum monoclonal gammaglobulin (M protein) level ≥ 5 g/L; or urinary M protein level ≥ 200 mg/24 hours; or serum immunoglobulin free light chain ≥ 100 mg/L (10 mg/dL) and abnormal serum immunoglobulin kap/lam light chain ratio.
3. Diagnosis of refractory/relapsed multiple myeloma: (1) Relapse is defined as the progression of disease after an initial response (≥MR) to prior therapy 60 days after cessation of therapy. (2) Refractory disease is defined as a <25% reduction in M protein or disease progression during treatment or within 60 days of stopping treatment.
4. ECOG assessment of 0, 1, or 2.
5. Life expectancy of at least 3 months.
6. The patient/legal guardian must be able to read, understand, and sign the informed consent form (ICF).

Exclusion Criteria:

1. Patient who currently participating or planning to participate in any interventional clinical study.
2. The investigator considers the patient unsuitable for participation in this study.
3. Non-secretory myeloma.
4. Subjects have received antimyeloma therapy within 2 weeks or 5 pharmacokinetic half-lives, whichever is longer, prior to initiation of treatment. This includes subjects who received a cumulative dose of corticosteroids greater than or equal to a 140 mg prednisone equivalent dose or a single dose of corticosteroids greater than or equal to a 40 mg/day dexamethasone equivalent dose within 2 weeks prior to initiation of treatment.
5. Subjects who have previously received an allogeneic stem cell transplant within 1 year prior to the date of enrollment and have not used immunosuppressive medications within 1 month prior to the date of enrollment.
6. Inadequate bone marrow reserve as defined by a platelet count <30 x 109/L or absolute neutrophil count <1.0 x 109/L.
7. Subject has clinically significant lung disease, including: (1) Subject has chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Please note that patients suspected of having COPD will be required to undergo FEV1 testing and subjects must be excluded if FEV1 is <50% of predicted normal. (2) Subjects who have had moderate or severe persistent asthma within the past 2 years or currently have any category of uncontrolled asthma. (Please note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma may participate in this study)
8. Subjects with clinically significant cardiac disease, including (1) Myocardial infarction within 6 months prior to Day 1 of Cycle 1, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina pectoris, congestive heart failure, New York Heart Association Class III-IV). (2) Cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE], 4th Edition, Grade 4 edition grade 2 or higher) or clinically significant ECG abnormalities. (3) Screening 12-lead ECG showing a baseline QT interval (QTcF) corrected by the Friedreichian formula >470 ms.
9. Severe hepatic dysfunction (total bilirubin 3 times normal or transaminases 3 times normal) unless associated with myeloma.
10. Creatinine clearance <20 mL/min.
11. Known allergy to components of the test product, or severe allergy or hypersensitivity to humanized products.
12. The subject has a concurrent serious and/or uncontrolled medical condition (e.g., uncontrolled diabetes mellitus, infections, hypertension, etc.) that may interfere with the study procedures or results or that, in the opinion of the investigator, may pose a risk to participation in this study.
13. Subjects known to be seropositive for human immunodeficiency virus (HIV) or have active hepatitis B or C.
14. History of active malignancy within the past 5 years, except squamous and basal cell carcinoma of the skin and carcinoma in situ of the cervix, or cured within 5 years with minimal risk of recurrence in the opinion of the local investigator, in agreement with the principal investigator.
15. Subjects known or suspected of not being able to comply with the study protocol (e.g. due to alcoholism, drug dependence, or psychological disorders), or the subject has any condition that, in the investigator's belief that participation would not be in the subject's best interest (e.g., detrimental to their well-being) or would likely prevent, limit, or confound protocol-specified assessments.
16. Pregnant or lactating females.
17. Peripheral neuritis ≥ grade 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 26 months
  Defined as the proportion of subjects who achieve stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) according to the 2016 International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Complete response rate (CR) | Up to 26 months
  Defined as the proportion of subjects whose serum and urine immunofixation electrophoresis are negative, and there is no soft tissue plasma cell tumor, with bone marrow plasma cells<5% by the 2016 International Myeloma Working Group (IMWG) criteria.
Progression free survival (PFS) | Up to 26 months
  PFS was defined as the time from the date of treatment initiation until the date of first documentation of definitive disease progression (PD) or date of death from any cause, whichever occurs first.
Overall survival (OS) | Up to 26 months
  OS will be measured from the date of registration to the date of the event (i.e., death) or the date of last follow-up to evaluate that event. Patients who are event-free at their last follow-up evaluation will be censored at that time point.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijuan Lin, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No